CLINICAL TRIAL: NCT06264856
Title: Flexible-bronchoscopy Trial for Moderate and Severe Thoracic Trauma Patients Without Brain Injury
Brief Title: Bronchoscopy for Thoracic Trauma Patients
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: The principal investigator will be studying abroad for one year. The study is expected to resume enrollment from December 1, 2024.
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 202210096RIND
Record Dates: First submitted 2023-04-03; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2023-04

CONDITIONS: Chest Trauma
MeSH Terms: conditions — Thoracic Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- bronchoscopic suction (Experimental): Bronchoscopic suction is a medical procedure used to remove excess mucus, secretions, and foreign objects from the airways through a bronchoscope. The patient would receive bronchoscopic sputum suction every 24-48 hrs after randomization until leaving ICU.. The patient could still receive blind negative pressure aspiration suction as the usual medical routine(every 2-4 hrs sputum suction if needed).
  Interventions: Procedure: bronchoscopic sputum suction
- blind negative pressure aspiration suction (Active Comparator): Negative pressure aspiration suction is a medical procedure that uses suction to remove fluids, mucus, or other materials from the body by creating a negative pressure or vacuum. The procedure involves inserting a catheter into the airway and applying negative pressure to the catheter to suction out the secretions or fluids. The patient would receive blind negative pressure aspiration suction as the usual medical routine(every 2-4 hrs sputum suction if needed).
  Interventions: Procedure: negative pressure aspiration suction

INTERVENTIONS:
Procedure: bronchoscopic sputum suction — Bronchoscopy is a medical procedure in which a flexible tube called a bronchoscope is passed through the mouth or nose and into the lungs. Bronchoscopic suction is a technique used during bronchoscopy to remove secretions, mucus, or foreign objects from the airways.
  The bronchoscope is equipped with a suction port and a suction channel that allows the doctor to remove fluids or other material from the airways. The suction port is connected to a vacuum source, and the suction channel runs through the bronchoscope and terminates at the tip of the instrument.
  Arms: bronchoscopic suction
Procedure: negative pressure aspiration suction — The procedure involves inserting a catheter into the airway and applying negative pressure to the catheter to suction out the secretions or fluids. The patient could receive sputum suction as medical routine (every 2-4 hrs) if needed.
  Arms: blind negative pressure aspiration suction

SUMMARY:
The study aims to evaluate the effectiveness of bronchoscopic sputum suction in patients with severe thoracic illness-induced respiratory failure. The study will compare the outcomes of patients who receive bronchoscopic sputum suction versus blind negative pressure aspiration for sputum removal. The study will measure baseline data, postoperative blood gas conditions, and clinical parameters, such as time of invasive ventilation, total time of ventilation, hospital stay, weaning success rate, reintubation rate, ventilator-associated pneumonia incidence, and fatality rate. The study aims to determine whether bronchoscopy-assisted sputum removal is superior to blind negative pressure aspiration in improving patient outcomes.

DETAILED DESCRIPTION:
The aim of the present randomized control trial is to assess the value of bronchoscopic sputum suction in patients with severe thoracic illness-induced respiratory failure. To decrease group differences in baseline characteristics and blood gas conditions, patients will be randomly assigned to receive either bronchoscopy-assisted or negative pressure aspiration for sputum suction, while the remaining treatment course will be the same. The study will measure major clinical indicators such as time of invasive ventilation, total time of ventilation, hospital stay, weaning success rate, reintubation rate, ventilator-associated pneumonia incidence, and fatality rate to provide strong evidence for the efficacy of each suction method.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be 20 years of age or older.
* Participants of all genders are eligible.
* Participants who are not in good health are not eligible.
* Participants with an Injury Severity Score greater than 9 and who have chest trauma are eligible.

Exclusion Criteria:

* Patients with traumatic brain injury.
* Patients with active pulmonary tuberculosis or other respiratory diseases with suspected contagion.
* Patients with poor blood clotting function or a tendency to bleed.
* Patients with aortic aneurysm. Patients with unstable vital signs or those who cannot maintain oxygen saturation above 90% while performing the test with Fraction of Inspired Oxygen (FiO2) greater than 80% or on 100% oxygen.
* Immunocompromised patients.
* Patients with acute massive hemoptysis.
* Patients with pre-existing neuromuscular diseases or those at high risk for arrhythmias, myocardial ischemia, or pulmonary embolism.
* Patients who are unable to clearly express their willingness to sign the informed consent form.
* Patients who have frequent intermittent sputum suction or are unable to fast for 4 hours due to their medical condition.

Ages: 20 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of pneumonia | 30 days after randomization
  diagnosis of pneumonia was determined according to radiologic evidence of new or progressive infiltrate of more than 48 hours and laboratory detection of a causative agent.
  The management and diagnosis of all patients was performed by a trauma specialist.

SECONDARY OUTCOMES:
Intensive Care Unit admission interval | 30 days
  measure the time of total Intensive Care Unit admission interval
admission interval | up to 24 weeks (from randomization to discharge)
  measure the time of total admission interval
tracheostomy rate | up to 24 weeks (from randomization to discharge)
  measure the rate of patient who receive tracheostomy in this admission
intubation rate | 90 days
  measure the rate of intubation rate

CONTACTS AND LOCATIONS:
Overall Officials: Hsien-Chi Liao, MD, Principal Investigator — Department of Traumatology, National Taiwain University Hospital
Locations (2):
- Taiwan (2):
  - Department of Traumatology, National Taiwain University Hospital, Taipei
  - NTUH Hsin-Chu Branch; NTUH Yun-Lin Branch, Taipei